CLINICAL TRIAL: NCT00586937
Title: Quality of Life in Lung Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-057
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer Survivors
Keywords: Lung Cancer Survivors
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Lung Cancer Survivors
  Interventions: Behavioral: questionnaires or telephone interview

INTERVENTIONS:
Behavioral: questionnaires or telephone interview — In the first phase, a random sample of lung cancer survivors will complete a comprehensive telephone interview or questionnaire by self-report focusing on assessment of quality of life and related covariates. We estimate the total time for completion of the survey by telephone interview or self-report to be 45-60 minutes. second phase of the study, a subset of telephone survey participants will take part in a focus group discussion that will explore their perceptions of barriers for delivery of post-treatment medical and psychosocial follow-up care.

SUMMARY:
The purpose of this study is to find out about the quality of life of individuals who have been diagnosed and treated for lung cancer (lung cancer survivors). By quality of life, we mean how you are feeling about different aspects of your life, including your physical health, your emotional health, and your ability to carry out daily activities. We are interested in people's opinions about their quality of life, as well as the factors that affect their quality of life. Learning about quality of life will help us to develop new services for lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Stage IA or IB NSCLC;
* Underwent surgical resection for NSCLC at MSKCC;
* From 1 to 5 years and 11 months post-treatment for NSCLC prior to study recruitment;
* No evidence of disease (NED) at the time of recruitment;
* Can be reached by telephone;
* Able to provide informed consent.

Exclusion Criteria:

* Undergoing active antineoplastic treatment;
* Major psychopathology or cognitive impairment likely in the judgment of the investigator to interfere with participation and compliance with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thoracic Surgery Database
Sampling Method: Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
To describe the health-related quality of life (HQOL) of lung cancer survivors and compare their HQOL with age- and gender-appropriate, population-based normative data. | 2 years

SECONDARY OUTCOMES:
To describe and identify covariates of HQOL in lung cancer survivors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org